CLINICAL TRIAL: NCT06062394
Title: Reducing Atherosclerotic Cardiovascular Disease (ASCVD) Through a Comprehensive Heart Disease Prevention Program (HDPP)
Brief Title: Penn Medicine Healthy Heart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 851832
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hypertension; Hyperlipidemias
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): This group will not receive the intervention and will continue with usual care.
- Penn Med Healthy Heart Program (Experimental): The Intervention group will receive the blood pressure monitor and move through the 4 HDPP modules of the intervention.
  Interventions: Behavioral: Penn Med Healthy Heart Program

INTERVENTIONS:
Behavioral: Penn Med Healthy Heart Program — Patients randomized to the intervention arm will be assigned a Patient Navigator (Clinical Research Coordinators, with support from Nurse Practitioners and a Medical Director) who will conduct an initial assessment with the patient to determine their main barriers to improving blood pressure and cholesterol control. The Patient Navigators will provide the patient with a home blood pressure cuff for remote monitoring, support from Way to Health text message reminders, referrals to established Penn Medicine smoking cessation programs, and referrals to nutrition and social workers as applicable. The Patient Navigators will help move the patients through four modules: Blood Pressure, Food Insecurity/Nutrition Screening, Statins, and Smoking Cessation. These modules provide patients with the chance to work on blood pressure, cholesterol control, access nutrition resources, and smoking cessation simultaneously or sequentially.
  Other Names: PMHH; HDPP
  Arms: Penn Med Healthy Heart Program

SUMMARY:
To leverage access to patients across the primary care network, EPIC tools for identifying eligible patients, and the Way to Health platform to launch and enroll a program that will be evaluated in a clinical trial that is focused on changing patient behavior and powered to detect differences in improving blood pressure and cholesterol over 6 months for Penn Medicine patients in West/Southwest Philadelphia and Lancaster.

DETAILED DESCRIPTION:
To leverage access to patients across the primary care network, EPIC tools for identifying eligible patients, and the Way to Health platform to launch and enroll Penn Medicine primary care patients into the Penn Medicine Healthy Heart, a six-month program for reduction of hypertension and hypercholesterolemia grounded in behavioral economics insights to increase uptake of and adherence to evidence-based interventions to reduce ASCVD risk. Penn Medicine Healthy Heart emphasizes proactive outreach and prevention outside of a traditional visit model using data assets to identify and risk stratify patients. The program aims to relieve overburdened PCPs through automated hovering technology coupled with a centralized, leveraged team of non-clinical navigators and nurse practitioners. The clinical trial will assess Penn Medicine Healthy Heart and will be powered to detect differences in improving blood pressure and cholesterol over 6 months for Penn Medicine patients in West/Southwest/Downtown Philadelphia and Lancaster, PA.

ELIGIBILITY:
Inclusion Criteria:

* On the Penn Medicine Primary Care Service Line registry
* Last 2 Blood Pressure readings with Systolic Blood Pressure >=140 from any outpatient encounter in the last 12 months AND
* ASCVD dx OR ASCVD risk score ≥10% OR Diabetes dx OR A1c ≥6.5 in last year OR Diabetes registry OR Last LDL ≥190 in past five years AND
* Not on a statinor PCSK9, Inclisiran OR on a Low-intensity/moderate-intensity statin) with LDL >100

Exclusion Criteria:

* Patients on PCSK9 inhibitors
* Documented statin allergy/ or intolerance in the EMR
* Pregnancy
* Breast feeding
* Markedly shortened life expectancy including:

  1. metastatic cancer
  2. hospice
  3. End Stage Renal Disease
  4. Congestive Heart Failure
  5. Dementia
* Is a non-English speaker requiring a translator
* Patients who do not have a cell phone

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1980 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Difference in mean Systolic Blood Pressure (SBP) | 6-month period
  Whether mean SBP is improved among those assigned to intervention vs those assigned to control
Difference in mean LDL-c | 6-month period
  Whether mean LDL-c is improved among those assigned to intervention vs those assigned to control

SECONDARY OUTCOMES:
Engagement in the BP intervention | 6-month period
  Engagement in the BP intervention as measured by number of participants who agree to receive blood pressure monitor
Difference in Diastolic Blood Pressure (DBP) | 6-month period
  Whether mean DBP is improved among those assigned to intervention vs those assigned to control Whether mean SBP is improved among those assigned to intervention vs those assigned to control

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Volpp KG, Mahraj K, Norton LA, Asch DA, Glanz K, Mehta SJ, Balasta M, Kellum W, Wood J, Russell LB, Fanaroff AC, Bakshi S, Jacoby D, Cohen JB, Press MJ, Clark K, Zhu J, Rareside C, Ashcraft LE, Snider C, Putt ME. Design and rationale of penn medicine healthy heart, a randomized trial of effectiveness of a centrally organized approach to blood pressure and cholesterol improvement among patients at elevated risk of atherosclerotic cardiovascular disease. Am Heart J. 2024 Dec;278:208-222. doi: 10.1016/j.ahj.2024.09.029. Epub 2024 Sep 27. PMID 39341482